CLINICAL TRIAL: NCT05511363
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Relapse Prevention Study to Evaluate the Safety and Efficacy of KarXT for the Treatment of Psychosis Associated With Alzheimer's Disease
Brief Title: A Study to Assess Efficacy and Safety of KarXT for the Treatment of Psychosis Associated With Alzheimer's Disease (ADEPT-1)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN012-0026; CN012-0026 (Other: Bristol-Myers Squibb Protocol ID); KAR-031 (Other: Karuna Pharmaceuticals Protocol ID)
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Psychosis Associated With Alzheimer's Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT (Experimental): Xanomeline and Trospium Chloride Capsules
  Interventions: Drug: KarXT
- Placebo (Placebo Comparator): Placebo Capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KarXT — KarXT 20 mg/2 mg TID KarXT 30 mg/3 mg TID KarXT 40 mg/4 mg TID KarXT 50 mg/5 mg TID KarXT 66.7/6.67 mg TID
  Arms: KarXT
Drug: Placebo — Placebo Capsules
  Arms: Placebo

SUMMARY:
This is a Phase 3, 38-week, randomized, double-blind, placebo-controlled, multicenter, outpatient study in subjects with psychosis associated with Alzheimer's Disease.

The primary objective of the study is to evaluate relapse prevention in subjects with psychosis associated with Alzheimer's Disease treated with KarXT compared to placebo. The secondary objectives of the study are to evaluate the time from randomization to discontinuation for any reason and safety and tolerability in subjects with psychosis associated with Alzheimer's Disease treated with KarXT compared to placebo.

ELIGIBILITY:
Inclusion Criteria

1. Is aged 55 to 90 years, inclusive, at Screening
2. Can understand the nature of the study and protocol requirements and provide a signed informed consent form before any study assessments are performed. If the subject is deemed not competent to provide consent, the following requirements for consent must be met.

   1. The subject's legally acceptable representative or caregiver/study partner, if local regulations allow, must provide informed consent
   2. The subject must provide informed assent
3. Meets clinical criteria for possible or probable Alzheimer's Disease
4. Has a Magnetic Resonance Imaging (MRI) or Computed Tomography (CT) scan of the brain (completed within the past 5 years) taken during or subsequent to the onset of dementia to rule out other central nervous system (CNS) disease that could account for the dementia syndrome. If not available, a non-contrast brain MRI or non-contrast head CT must be done during screening.
5. Living at the same home or residential assisted-living facility for a minimum of six weeks before Screening
6. Capable of self-locomotion (alone or with the aid of an assistive device) and have an identified or proxy caregiver (spends approximately 10 hours/week with the subject) that is willing to:

   1. Attend all visits and report on subject's status
   2. Oversee subject compliance with medication and study procedures
   3. Participate in the study assessments and provide informed consent to participate in the study
7. History of psychotic symptoms (meeting International Psychogeriatric Association [IPA] criteria) for at least 2 months prior to Screening.
8. Clinical Global Impressions-Severity (CGI-S) scale with a score ≥4 (moderate) at Screening and Baseline. CGI-S requires the assessor to consider aspects of the psychosis prior to providing a global assessment of severity. These aspects include hallucinations and delusions.
9. Subjects are required to meet at least one of the following criteria at Screening and Baseline:

   1. Moderate to severe delusions, defined as Neuropsychiatric Inventory-Clinician (NPI-C): Delusions domain score of ≥2 on two of the eight items OR
   2. Moderate to severe hallucinations, defined as NPI-C: Hallucinations domain score of ≥ 2 on two of the seven items.
10. Mini-Mental State Examination (MMSE) score of 8 to 22, inclusive, at Screening
11. If the subject is taking a cholinesterase inhibitor and/or memantine, they must have been on a stable dose for 6 weeks prior to Screening and be willing to maintain a stable dose for the duration of the study.
12. Subject is willing and able to visit the clinic in an outpatient setting for the study duration, follow instructions, and comply with the protocol requirements
13. BMI must be within 18 to 40 kg/m2 inclusive
14. Female subjects must not be pregnant or breastfeeding. Women of childbearing potential (WOCBP), or men whose sexual partners are WOCBP, must be able and willing to use at least 1 highly effective method of contraception during the study and for at least 1 menstrual cycle (e.g., 30 days) after the last dose of IMP or matching placebo. Sperm donation is not allowed for 30 days after the final dose of the IMP or matching placebo.

Exclusion Criteria

1. Psychotic symptoms that are primarily attributable to a condition other than the Alzheimer's Disease causing dementia
2. History of major depressive episode with psychotic features during the 12 months prior to Screening
3. History of a diagnosis of bipolar disorder, schizophrenia, or schizoaffective disorder
4. Significant or severe medical conditions including pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, cardiovascular or oncologic disease, or any other condition that, in the opinion of the Investigator, could jeopardize the safety of the subject, ability to complete or comply with the study procedures or validity of the study results
5. Significant or severe renal impairment based on a screening cutoff for Estimated Glomerular Filtration Rate (eGFR) of <60 mL/min/1.73 m2
6. History of ischemic stroke within 12 months prior to Screening or any evidence of hemorrhagic stroke
7. History of cerebral amyloid angiopathy, epilepsy, central nervous system neoplasm, unstable thyroid function, or unexplained syncope
8. Any of the following:

   1. New York Heart Association Class 2 congestive heart failure
   2. Grade 2 or greater angina pectoris
   3. Sustained ventricular tachycardia
   4. Ventricular fibrillation
   5. Torsade de pointes
   6. Implantable cardiac defibrillator
9. Myocardial infarction within the 6 months prior to Screening
10. Personal or family history of symptoms of long QT syndrome as evaluated by the investigator
11. Human immunodeficiency virus, cirrhosis, biliary duct abnormalities, hepatobiliary carcinoma, and/or active hepatic viral infections as indicated by medical history or liver function tests results
12. History or high risk of urinary retention, gastric retention, or narrow-angle glaucoma as evaluated by the investigator
13. For males only, any one of the following:

    1. History of bladder stones
    2. History of recurrent urinary tract infections
    3. Serum prostate specific antigen (PSA) > 10 ng/mL at Screening
    4. An International Prostate Symptom Score (IPSS) of 5 (almost always) on items 1, 3, 5, or 6
    5. A sum of scores on IPSS items 1, 3, 5, and 6 of ≥9
14. History of irritable bowel syndrome (with or without constipation) or serious constipation requiring treatment within the last 6 months
15. Risk of suicidal behavior during the study as determined by clinical assessment and/ or C-SSRS
16. Clinically significant abnormal finding on the physical examination, electrocardiogram, or clinical laboratory results at Screening
17. Urine toxicology screen is positive substances other than cannabis or benzodiazepines (both cannabis and short-or medium-acting benzodiazepines are allowed in limited quantities during the study) unless approval has been given by the Medical Monitor
18. Recent history of receiving monoamine oxidase inhibitors, anticonvulsants (e.g., lamotrigine, divalproex), lithium, tricyclic antidepressants (e.g., imipramine, desipramine), or any other psychoactive medications except for as-needed anxiolytics (e.g., lorazepam, chloral hydrate)

    1. Selective serotonin reuptake inhibitors and serotonin norepinephrine reuptake inhibitors taken at a stable dose for at least 8 weeks prior to Screening may be permitted
    2. Mirtazapine or trazodone may be used as a hypnotic if started at least 8 weeks prior to Screening. If needed, an extension (up to two weeks) of the Screening Period may be allowed with approval of the Sponsor/Medical Monitor.
19. If, in the opinion of the Investigator and/or Sponsor/Medical Monitor, subject is unsuitable for enrollment in the study or subject has any finding that, in the view of the Investigator and/or Sponsor/ Medical Monitor, may compromise the safety of the subject or affect his/her ability to adhere to the protocol visit schedule or fulfill visit requirements
20. Positive test for coronavirus (COVID-19) within 2 weeks before or at Screening; antigen or PCR local testing can be done at the discretion of the Investigator
21. Unable to taper and discontinue a concomitant medication that would preclude participation in the study
22. Prior exposure to KarXT
23. Experienced any significant adverse events due to trospium, including a known hypersensitivity to trospium
24. Participation in another clinical study in which the subject received an experimental or investigational drug within 3 months before Screening or has participated in more than 2 clinical studies in the past year

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to relapse during the 38-week study | Week 38

SECONDARY OUTCOMES:
Time from randomization to discontinuation for any reason during the 38-week study | Week 38

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (113):
- United States (58):
  - Local Institution - 1029, Homewood, Alabama
  - Local Institution - 1044, Phoenix, Arizona
  - Local Institution - 1033, Encino, California
  - Local Institution - 1031, Irvine, California
  - ATP Clinical Research-302 W La Veta Ave, Orange, California
  - Local Institution - 1043, Pasadena, California
  - Local Institution - 1047, San Marcos, California
  - Sunwise Clinical Research, LLC - Walnut Creek - IVY - PPDS, Walnut Creek, California
  - Local Institution - 1014, Colorado Springs, Colorado
  - Local Institution - 1013, Stamford, Connecticut
  - Local Institution - 1011, Boca Raton, Florida
  - Envision Trials LLC, Bonita Springs, Florida
  - Local Institution - 1015, Bradenton, Florida
  - K2 Medical Research - Winter Garden, Clermont, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Local Institution - 1045, Doral, Florida
  - Local Institution - 1046, Hialeah, Florida
  - Local Institution - 1024, Hialeah, Florida
  - Local Institution - 1052, Hialeah, Florida
  - Local Institution - 1049, Homestead, Florida
  - K2 Medical Research - Maitland, Maitland, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - Local Institution - 1005, Miami, Florida
  - Floridian Neuroscience Institute-1901 SW 1 St, Miami, Florida
  - Local Institution - 1010, Miami, Florida
  - Local Institution - 1143, Miami, Florida
  - Local Institution - 1009, Miami, Florida
  - Future Care Solution LLC, Miami, Florida
  - South Florida Research Phase I-IV, Inc. - Miami, Miami, Florida
  - Novel Clinical Research Center, LLC., Miami, Florida
  - Local Institution - 1111, Miami, Florida
  - Coral Research Clinic & Coral Diagnostic Center, Miami, Florida
  - Local Institution - 1042, Miami, Florida
  - Local Institution - 1032, Miami Lakes, Florida
  - Local Institution - 1026, Miami Springs, Florida
  - Local Institution - 1027, Ocala, Florida
  - Local Institution - 1012, Pensacola, Florida
  - Local Institution - 1008, St. Petersburg, Florida
  - Local Institution - 1050, Tampa, Florida
  - K2 Medical Research - Tampa, Tampa, Florida
  - Local Institution - 1040, The Villages, Florida
  - Local Institution - 1037, Chicago, Illinois
  - Local Institution - 1018, Manhasset, New York
  - Local Institution - 1030, New York, New York
  - Local Institution - 1051, New York, New York
  - Local Institution - 1017, New York, New York
  - Local Institution - 1002, Staten Island, New York
  - Local Institution - 1034, Stony Brook, New York
  - Five Towns Neurology, PC, Woodmere, New York
  - Local Institution - 1003, Canton, Ohio
  - Local Institution - 1028, Oklahoma City, Oklahoma
  - Local Institution - 1016, Oklahoma City, Oklahoma
  - Local Institution - 1019, Allentown, Pennsylvania
  - Local Institution - 1035, Charleston, South Carolina
  - Local Institution - 1038, Franklin, Tennessee
  - Local Institution - 1022, Flower Mound, Texas
  - Local Institution - 1036, Frisco, Texas
  - Clinical Trial Network - 7080 Southwest Fwy, Houston, Texas
- Bulgaria (5):
  - Medical Center Sveti Naum EOOD, Sofia, Sofia-Grad
  - Local Institution - 4505, Sofia, Sofia-Grad
  - Local Institution - 4502, Sofia, Sofia-Grad
  - Medical Center Medconsult Pleven OOD, Pleven
  - Local Institution - 4504, Vratsa
- Croatia (5):
  - Local Institution - 4102, Zagreb, City of Zagreb
  - Local Institution - 4103, Zagreb, City of Zagreb
  - Local Institution - 4105, Zagreb, City of Zagreb
  - Klinika za psihijatriju Vrapce, Zagreb, City of Zagreb
  - Psychiatric Clinic Sveti Ivan, Zagreb, City of Zagreb
- Czechia (6):
  - CLINTRIAL s.r.o., Prague, Praha, Hlavní Mesto
  - Local Institution - 4003, Brno, South Moravian
  - Neuroterapie KH, s.r.o, Kutná Hora
  - A-SHINE s.r.o., Pilsen
  - Clinoxus s.r.o., Prague
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
- France (3):
  - Local Institution - 2501, Reims, Marne
  - Local Institution - 2502, Dijon
  - Local Institution - 2503, Rouen
- Germany (3):
  - Local Institution - 2401, Böblingen, Baden-Wurttemberg
  - Local Institution - 2403, Bayreuth, Bavaria
  - Local Institution - 2402, Homburg, Saarland
- Italy (9):
  - Local Institution - 2301, Rome, Lazio
  - Local Institution - 2306, Baggiovara, Modena
  - Local Institution - 2307, Ponderano (Biella), Piedmont
  - Local Institution - 2308, Florence, Tuscany
  - Local Institution - 2304, Milan
  - Local Institution - 2305, Monza
  - Local Institution - 2302, Pisa
  - Local Institution - 2303, Roma
  - Local Institution - 2309, Roma
- Serbia (8):
  - University Clinical Center of Serbia - Pasterova 2 - PPDS, Belgrade, Belgrade
  - Clinical Hospital Center Dragisa Misovic Dedinje, Belgrade
  - Local Institution - 4307, Belgrade
  - Military Medical Academy, Belgrade
  - Special Hospital for Psychiatric Diseases Kovin, Kovin
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Centre of Vojvodina, Novi Sad
  - Local Institution - 4311, Vršac
- Slovakia (6):
  - Univerzitna nemocnica L Pasteura Kosice-Rastislavova 43, Košice, Košice Region
  - MUDr. Beata Dupejova, Neurologicka ambulancia, s.r.o., Banská Bystrica
  - KONZILIUM s.r.o, Dubnica nad Váhom
  - EPAMED s.r.o, Košice
  - Crystal Comfort, s.r.o., Vranov nad Topľou
  - Local Institution - 4404, Žilina
- Spain (7):
  - Local Institution - 2205, Barcelona
  - Local Institution - 2207, Madrid
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Hospital Victoria Eugenia, Seville
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Provincial de Zamora, Zamora
  - Hospital Viamed Montecanal, Zaragoza
- United Kingdom (3):
  - Local Institution - 2103, Swindon, Wiltshire
  - Local Institution - 2105, Aberdeen
  - Local Institution - 2104, Motherwell

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05511363.html